CLINICAL TRIAL: NCT05084612
Title: Comparison Between a Two Person Insertion With Lateral Rotation Technique of Laryngeal Mask Airway and the Classic Technique; a Randomized Controlled Trial
Brief Title: Comparison Between a Two Person Insertion With Lateral Rotation Technique of LMA and the Classic Technique
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The 107 the principal investigator was changed on November, 2022.
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC4-4-2021
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (S) (Placebo Comparator): LMA will be placed using the standard Brain's insertion technique.
  Interventions: Device: standard LMA insertion
- Rotational group (R) (Active Comparator): LMA will be placed using a two Person Insertion with lateral rotation technique.
  Interventions: Device: New technique LMA insertion

INTERVENTIONS:
Device: standard LMA insertion — Following pre-oxygenation, anaesthesia will be induced with atropine 0.1mg/kg, Fentanyl 2 µg /kg, Propofol 2 mg/kg and atracurium 0.5 mg/kg. When neuromuscular blockade will be complete
  the laryngeal mask will be inserted with using the standard method described by Brain; after lubrication of the posterior aspect of the partially deflated mask, the patient's head will be positioned with head extended at the atlanto-axial joint and flexed at the neck with non-dominant hand. The LMA will be held like a pen and index finger will be placed at the junction of LMA tube and cuff. Index finger will be used to press the LMA against hard palate and posterior pharyngeal wall until definite resistance felt at the base of the hypopharynx. LMA will then be held with non-dominant hand and index finger will be removed.
  Arms: control group (S)
Device: New technique LMA insertion — Following pre-oxygenation, anaesthesia will be induced with atropine 0.1mg/kg, Fentanyl 2 µg /kg, Propofol 2 mg/kg and atracurium 0.5 mg/kg. When neuromuscular blockade will be complete LMA will be inserted by a two Person Insertion with lateral rotation Technique; after lubrication of the posterior aspect of the partially deflated mask, the assistant will achieve jaw thrust and mouth opening then LMA will be inserted by the anaesthiologist. LMA will be inserted by holding the mask by index, middle finger and thumb; after insertion of the entire cuff inside the mouth, the LMA will be rotated anticlockwise through 90° (the inner surface of LMA will be directed medially towards the mouth cavity) and advanced through the side of the tongue until resistance felt, then turned back in the hypopharynx.
  Arms: Rotational group (R)

SUMMARY:
The laryngeal Mask Airway was developed by Brain in 1981 and was available for clinical use in the United States by 1992 and has become very popular in routine medicine practice during 10 past years . LMA would serve as a choice to be used in the emergency situations even by the inexperienced users . Nowadays due to the increasing number of outpatient anesthesia and use of short-acting anesthetics almost without the use of any muscle relaxants requires an appropriate way for safe LMA insertion. As LMA insertion is generally performed blindly, clinicians are always in search of how to place and maintain the LMA in appropriate position.

DETAILED DESCRIPTION:
The standard method of insertion described by Dr. Brain is relatively easy, but sometimes it is impossible to insert the LMA with the standard method. However ease and time of airway management may be of special importance in emergent situations. Since its inception the LMA has undergone various modifications in type and material, which have made other methods of insertion possible, quicker and easier than the standard method. Intraoral manipulation can put the operator at risk of finger trauma and infection. However it is not possible to avoid intraoral manipulation when the standard technique or the classic LMA is used.

Therefore, many studies were seeking to find new methods to improve this technique. Hwang et al. first described The 90° rotation technique in adults that involves the following steps: the entire cuff of the LMA is inserted inside the mouth, rotated counter-clockwise through 90° and advanced until the resistance of the hypopharynx is felt . The use of this method is known to increase the success rate of insertion and decrease the incidence of blood staining of the LMA and sore throat compared to standard technique . Ghai et al. showed that rotational technique may be considered as the first technique of choice for classical laryngeal mask airway insertion in children . Lopez-Gil and colleagues reported a decrease in complications with the increase in the skill of the anaesthetist . PARVIZ et al. described a two person technique which performed by the technician who performs mouth opening and jaw thrust and the anesthesiologist who inserts the laryngeal mask. They considered it as a safe and effective method to establish a secure airway in anesthetized patients.. other studies have shown that LMA insertion with partially inflated cuff is easier than deflated cuff .

Current study will combine two methods of LMA insertion including two-persons and lateral rotational techniques and compare them with the standard insertion method regarding the success rate and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status grade I-II,
* Age between 20-55 years old
* undergoing minor surgeries under general anaesthesia using LMA

Exclusion Criteria:

* patients at Risk of aspiration,
* Mouth opening ˂ 2.5 cm,
* BMI ≥ 35 kg/m2,
* dental problems,
* recent history of upper airway infection,
* gastro-oesophageal reflux disease and
* limited extension of the neck.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
the success rate of first attempt insertion of the LMA | from induction of anesthesia till patient connected to the ventilator.
  confirmed insertion of LMA without need for further attempts.

SECONDARY OUTCOMES:
LMA insertion time | up to 30 minutes post-induction of anesthesia
  the period from mouth passage of the device to effective ventilation after inflation of the cuff.
The number of insertion attempts | up to 30 minutes post-induction of anesthesia
  If ventilation is still ineffective, re-insertion will be tried up to three times. After third unsuccessful attempt then one attempt will be made using the alternative approach, if still unsuccessful endotracheal tube will be inserted.
number of manipulations needed during insertion | up to 30 minutes post-induction of anesthesia
  manipulations like jaw thrust, chin lift, and extension and flexion of the neck
The incidence of complications following insertion of LMA | up to 1 day postoperative
  including; laryngospasm, hypoxaemia (SpO2 < 90%) and trauma (assessed by blood stained LMA on removal)
Heart rate (HR) | first 15 minutes post-induction of anesthesia
  monitoring of stress response during the maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided